CLINICAL TRIAL: NCT06524609
Title: Clinical Study of EGCG for the Prevention and Treatment of Peripheral Neuropathy Induced by Taxane (TIPN)
Brief Title: EGCG for the Prevention and Treatment of TIPN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Han Xi Zhao (Other)
Collaborators: The Fourth People's Hospital of Jinan (Unknown)
Responsible Party: Sponsor-Investigator, Han Xi Zhao, chief physician, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGCG-TIPN
Record Dates: First submitted 2024-06-28; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: peripheral neurotoxicity; Chemotherapy-Induced Peripheral Neuropathy
MeSH Terms: interventions — epigallocatechin gallate; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGCG GROUP (Experimental): EGCG administration was initiated when Grade II CIPN occurred first time. EGCG solution is applied to the patient's hands/feet with a soft-bristled brush, approximately 0.05 ml/cm2. 3 times daily, and may be covered with film gloves/cling film for approximately 20-30 minutes after application. Use continuously for at least 1 week.
  Interventions: Drug: Epigallocatechin-3-Gallate
- CONTROL GROUP (Placebo Comparator): 75% alcohol
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Epigallocatechin-3-Gallate — After determining the optimal dose, the efficacy of EGCG was compared with that of a control group (75% alcohol).
  Arms: EGCG GROUP
Drug: Alcohol — After determining the optimal dose, the efficacy of EGCG was compared with that of a placebo control group (75% alcohol).
  Arms: CONTROL GROUP

SUMMARY:
Patients treated with paclitaxel analogs and experiencing Taxane-induced peripheral neurotoxicity (TIPN) of degree I or higher were treated with EGCG solution. The safety of topical EGCG solution for the treatment of TIPN and the optimal drug concentration were also verified by a phase I trial. The efficacy and safety of the optimal EGCG concentration obtained in the phase I trial were further analyzed in a randomized controlled phase II trial. Meanwhile, the predictive molecules of TIPN efficacy were initially explored by detecting patients' hematological related indexes. The optimal dose concentration, safety and efficacy of EGCG to ameliorate the neurotoxicity caused by paclitaxel-related drugs were clarified.

DETAILED DESCRIPTION:
Enrolled patients with tumors that developed CIPN of degree II or greater who received albumin-bound paclitaxel chemotherapy. The baseline degree of CIPN in patients was evaluated by CTCAE and TNS as well as the EORTC-CIPN20 scale. EGCG was purchased from HEP Biotech Co., Ltd (Ningbo, Zhejiang, China) and freshly dissolved in 75% alcohol by volume. EGCG concentrations were climbed from 1% according to the modified Fibonacci method for 4 dose groups. EGCG administration was initiated when Grade II CIPN occurred first time. EGCG solution is applied to the patient's hands/feet with a soft-bristled brush, approximately 0.05 ml/cm2. 3 times daily, and may be covered with film gloves/cling film for approximately 20-30 minutes after application. Use continuously for at least 1 week. By comparing and analyzing the degree of reduction in CECAE, TNS, and EORTC scale data before and after EGCG treatment in patients with degree II CIPN, the optimal EGCG drug dosing concentration was obtained to validate safety. The EGCG concentration obtained from the phase I trial was also used to prospectively conduct a randomized controlled phase II clinical trial to further validate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed cancer
* Received ≥1 cycle of systemic chemotherapy with albumin-bound paclitaxel
* Adequate hematologic, hepatic, and kidney function profile
* CIPN was evaluated by CTCAE as grade ≥2
* Urine or serum pregnancy test within 3 days prior to first dose in female subjects of childbearing potential
* Subjects were willing and able to comply with the schedule of visits, treatment protocols, laboratory tests, and compliance with other requirements of the study.

Exclusion Criteria:

* The presence of a pre-existing condition that may result in a high risk of neuropathy: diabetes mellitus, thyroid disease, prior treatment with other medications that may result in neurological damage, alcoholism, familial neuropathy
* Concurrent enrollment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study
* Have taken medication for the treatment or prevention of peripheral neuropathy in the 2 weeks prior to screening, or have received traditional Chinese medicine (acupuncture, moxibustion, herbal medicine, cupping) within 1 month
* Known active tuberculosis (TB): Subjects suspected of having active TB need to be excluded by clinical examination.
* Known active syphilis infection.
* Known allergy to any component of any study drug; including alcohol allergy.
* Known history of mental illness, drug dependence, alcoholism or drug addiction.
* Any pre-existing or current medical condition, treatment, or laboratory test abnormality that may confound the results of the study, interfere with the subject's ability to participate in the study in its entirety, or participation in the study may not be in the subject's best interest.
* Localized or systemic disease not due to malignancy; or disease or condition secondary to a tumor that may result in a higher medical risk and/or uncertainty in the evaluation of survival, such as tumor-like leukemic reaction (white blood cell count >20 x 109/L), malignant manifestations (e.g., known weight loss of more than 10% in the 3 months prior to Screening).
* Be pregnant or breastfeeding, or plan to breastfeed during the study. Other conditions that the investigator considers inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
sensory nerves and motor nerves of CTCAE | 42 days
  CTCAE（Common Terminology Criteria for Adverse Events）: A minimum of 1 grade and maximum of 5 grades.
TNS（Total Neuropathy Score） | 42 days
  TNS（Total Neuropathy Score）: Including sensory nerves, motor nerves and tendon reflexes, etc., 10 indicators, with a minimum of 1 grade and maximum of 5 grades each, and the scores of the 10 indicators were added together for a total.
EORTC Scale（European Organization for Research and Treatment of Cancer TIPN-specific Quality of Life Quality of Life Questionnaire for CIPN） | 42 days
  The scale consists of 9 scales for sensory, motor, and autonomic nerves, same grading and calculation method as the TNS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hanxi Zhao, Dr., Study Director — Institute of Radiation Medicine, Shandong First Medical University
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital (Shandong Academy of Medical Sciences), Jinan, Shandong, China